CLINICAL TRIAL: NCT07065396
Title: Virtual Reality and Cranial Nerve Neuromodulation in the Management of Chronic Pain in Veterans: a Pilot Study
Brief Title: Virtual Reality and Cranial Nerve Neuromodulation to Manage Chronic Pain
Acronym: VR & CN-NINM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Chronic Pain Center of Excellence for Canadian Veterans (Unknown); Quebec Pain Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-5448a
Record Dates: First submitted 2025-06-19; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; PTSD - Post Traumatic Stress Disorder
Keywords: Chronic pain; PTSD; Veterans; Autonomic nervous system; Virtual reality (VR); Cranial nerve non-invasive neuromodulation (CN-NINM)
MeSH Terms: conditions — Chronic Pain; Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study model is a factorial crossover study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality (VR) (Experimental): VR interventions (hypnotic suggestions with auditory and visual calming stimulations) will applied for 20 minutes.
  Interventions: Procedure: Virtual reality
- Virtual reality (VR) + Cranial nerve non-invasive neuromodulation (CN-NINM) (Experimental): CN-NINM will be applied during the VR interventions (20 min).
  Interventions: Procedure: Virtual reality; Procedure: Cranial nerve non-invasive neuromodulation (CN-NINM)
- Virtual reality (VR) + sham CN-NINM (Placebo Comparator): Sham CN-NINM (no stimulation) will be applied during the VR interventions (20 min).
  Interventions: Procedure: Virtual reality; Procedure: Placebo CN-NINM

INTERVENTIONS:
Procedure: Virtual reality — The VR intervention will take place in a quiet room. The participant will be installed in a seated position, wearing a virtual reality headset that includes an audio device playing sounds. The eyes are covered by a mask featuring a screen showing calming 3D VR images (e.g. beach landscapes), designed by our team. The intervention lasts 20 minutes. The hypnotic suggestions with auditory and visual calming stimulations will help the person to focus on the present moment, to reduce anxiety and painful sensations.
Procedure: Cranial nerve non-invasive neuromodulation (CN-NINM) — During each intervention including CN-NINM, this latter will be applied for 20 minutes, with the help of a portable stimulator comprising a network of 18 electrodes, directly on the tongue of the participants. The participants will hold the CN-NINM in place by pressing their tongue upwards. The CN-NINM will generate high-frequency pulses (50 µsec to 150 Hz), and the intensity of the stimulus will be set by each participant to a comfortable level of sensation, similar to the sensation in the mouth of a soft drink.
  Arms: Virtual reality (VR) + Cranial nerve non-invasive neuromodulation (CN-NINM)
Procedure: Placebo CN-NINM — In this study, we will have a control intervention which will be placebo CN-NINM. For placebo CN-NINM, participants will wear the device such as the real CN-NINM group, without having experienced the tingling sensation beforehand, so they will not know what the CN-NINM potential effect is.
  Arms: Virtual reality (VR) + sham CN-NINM

SUMMARY:
In Canada, veterans suffer from chronic pain at twice the rate of the general population. This pain is often linked to post-traumatic stress disorder (PTSD), and both have a major impact on their quality of life. The autonomic nervous system (ANS) plays a key role in these pathologies, making its modulation a promising therapeutic target. Virtual reality (VR) is already being used to alleviate pain and PTSD in veterans, mainly by modulating ANS reactivity. Two types of VR exist: prolonged exposure (desensitization) and the calming effect, the latter being better tolerated and more suitable for rebalancing the ANS. However, its effects on pain remain modest and temporary. To reinforce these benefits, it is proposed to combine VR with a new approach called cranial nerve non-invasive neuromodulation (CN-NINM), an innovative technique that allows the generation of a direct flow of neuronal impulses via the stimulation of the tongue. The goal of this project is therefore to document the efficacy of VR and the combination of VR and CN-NINM on pain and ANS in veterans suffering from chronic pain and PTSD. VR, CN-NINM and the combination of the two will be applied for 20 minutes. Clinical pain, experimental pain and ANS reactivity will be assessed before and after the interventions. At the end of this study, it is expected that the investigators will be able to document the type of effect CN-NINM could have, and that it could become a complementary therapeutic option.

DETAILED DESCRIPTION:
In Canada, many veterans suffer from chronic pain, with a prevalence twice as high as that of the general population. Chronic pain is often linked to post-traumatic stress disorder(PTSD). Together, these two conditions impact on the functioning and quality of life of veterans. Recent studies suggest that the autonomic nervous system (ANS) plays a central role in the pathophysiology of chronic pain and PTSD, making it a prime therapeutic target.

Virtual reality (VR) is already being used with veterans, and its effectiveness in relieving pain and PTSD is well documented in veterans, notably by modulating ANS reactivity. Two types of VR approaches are commonly used: VR with prolonged exposure (desensitization) and VR with a calming effect (aimed at normalizing the stress response and SNA reactivity).The latter is better tolerated than prolonged-exposure VR and remains better suited to rebalancing ANS reactivity and relieving symptoms. It calms the ANS and relieves pain (acute and chronic) when combined with traditional rehabilitation, but its effects on pain intensity remain modest and limited in time.

To optimize the benefits of VR, it is proposed to combine VR with a non-pharmacological method, as suggested by experts. This non-pharmacological approach is cranial nerve non-invasive neuromodulation (CN-NINM). CN-NINM is an innovative approach that stimulates the cranial nerves via electrodes placed directly on the tongue; the impulses reach and modulate the activity of ANS structures located in the brainstem. These structures are linked to autonomic functions and pain modulation. This combination could reinforce and prolong the positive effects of VR on veterans' pain.

Objectives: 1) To document the effect of VR (an intervention currently provided) on pain and ANS reactivity in veterans with PTSD, 2) to assess the ability of CN-NINM (vs sham CN-NINM) to potentiate the effects of VR on pain and on ANS reactivity.

Methods: In this within-subjects factorial crossover design, 15 veterans will be recruited. Sociodemographic, pain and PTSD-related variables will be collected to confirm participant eligibility. Prior to the interventions, participants will undergo an assessment of both clinical pain (intensity and unpleasantness of pain, numerical scale 0-10) and experimental pain. The tonic thermal experimental pain paradigm involves the application of a thermode (hotplate) to participants' forearms. Thermal nociceptive stimuli will be induced for 2 minutes on the participants' forearm using the thermode. Although the temperature remains constant for the entire 2 minutes, the participant will be informed that the temperature may increase, decrease, or remain stable during the procedure. The participant will then, at all times, evaluate the intensity of the pain with a visual analogue scale connected to a computer(CoVAS: visual analogue scale from 0 to 100).

Additionally, participants will complete clinical questionnaires assessing anxiety, pain and PTSD-related symptoms. Various autonomic measures (blood pressure, heart rate reactivity [HRV], electrodermal response) will also be taken to characterize ANS reactivity before and after each intervention. Participants will receive the 3 interventions (VR, VR+CN-NINM and VR+ sham CN-NINM) randomly assigned. The VR headset will broadcast calming images for 20 minutes. CN-NINM will be applied, using a portable stimulator, placed directly on the tongue of the participants for 20 minutes simultaneously with VR.

ELIGIBILITY:
Inclusion Criteria:

1. Be a veteran;
2. Be ≥30 years old;
3. Have a diagnosis of chronic musculoskeletal pain (pain > 6 months);
4. Have been diagnosed with PTSD by a health professional and/or have a PTSD Checklist for DSM-5 (PCL-5) score > 30/80 and
5. Speak English or French.

Exclusion Criteria:

1. Bipolar disorder, psychosis;
2. Neuropathic pain (based on the Neuropathic Pain Diagnosis and Questionnaire (DN4));
3. Visual disorders or photosensitivity, color blindness;
4. Epilepsy, motion sickness and
5. Any containdications to CN-NINM.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate for the project | Information will be assessed at the end of the recruitment period, at week 28
  This outcome will be compiled by the total number of participants recruited, divided by the average number of months recruiting.
Refusal to participate and the reasons | Information will be assessed throughout the project recruitment period (average of 7 months)
  Participant refusal will be quantified by recording the number of individuals who declined to take part in the study. The reasons for refusal will also be documented.
Dropped out rate of the project in percent | Information will be assessed through project completion, an average of 9 months
  The dropout rate will be determined by calculating the proportion of participants who discontinued their participation relative to the total number of participants initially enrolled, expressed as a percentage.
Adherence to the interventions (VR, VR + CN-NINM, VR + CN-NINM placebo) in percent | Information will be assessed through study completion, an average of 9 months
  Adherence to interventions will be calculated by the number of visits completed out of the total number expected X 100%, by attrition and loss to follow-up.
Safety-related informations for each intervention as assessed by a questionnaire | Information will be assessed through study completion, an average of 9 months
  Safety-related informations for each intervention will be assessed with a questionnaire that will provide a number and percentage of participants who have experienced adverse events (frequency, type and severity of adverse events).

SECONDARY OUTCOMES:
Change in pain intensity on the CoVAS | The assessments will be done at the baseline and just after the 20 minutes of application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo).
  Change in pain intensity will be calculated by the difference between the pain felt andreported on the CoVAS (average of the 2 minutes) before and after the 20 minutes of application of each intervention. The score on the CoVAS ranges between 0 (no pain) to 100 (maximal pain).
Change in measures of blood pressure | The assessments will be done at baseline, during the 20 min application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo) and just after the 20 min application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo).
  Change in measures of blood pressure will be assessed with NIBP100E Finger Cuff Sensors and Blood Pressure Cuff from BIOPAC.
Change in heart rate variability | The assessments will be done at the baseline, during the 20 minutes of application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo) and just after the 20 minutes of applications of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo).
  Change in heart rate variability will be assessed with ECG Electrocardiogram Amplifier (MP200) from BIOPAC.
  Investigators will look at:
  * Root Mean Square of Successive Differences or RMSSD (measurement that reflects the activity of the parasympathetic nervous system),
  * High Frequencies or HF (representing the activity of the parasympathetic nervous system) and
  * Low Frequencies/High Frequencies [LF/HF] ratio (indicator of the balance between the activity of the sympathetic nervous system (SNS) and the parasympathetic nervous system (SNP)).
Change in electrodermal response | The assessments will be done at the baseline, during the 20 min application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo) and just after the 20 min application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo).
  Change in electrodermal response will be assessed with the EDA finger transducer from BIOPAC.
Change in pain intensity and impact on physical function using the Brief Pain Inventory (BPI) | The questionnaire will be done at the baseline (T0), beginning and just after the 20 minutes of application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo) and one week after the last intervention.
  Change in pain intensity and impact will be assessed using a scored questionnaire. The questionnaire score is divided into two dimensions: the pain impact on physical function score (/70) and the severity score (/40). A high score would indicate severe pain with a significant impact on physical function.
Change in the qualitative aspect of pain with the McGill Pain Questionnaire (MPQ) | The questionnaire will be done at the baseline (T0), beginning and just after the 20 min application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo) and one week after the last intervention.
  Change in the qualitative aspect of pain will be measured with the McGill Pain Questionnaire, a scored multi-dimensional questionnaire. The questionnaire score range from 0 (no pain) to 78 (severe pain). A higher total score indicates a more intense pain experience.
Change in pain-related disability using the Pain Disability Questionnaire (PDQ) | The questionnaire will be done at the baseline (T0), beginning and just after the 20 min application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo) and one week after the last intervention.
  Change in pain-related disability will be evaluated using the PDQ. The total PDQ score range from 0 to 150. A high score indicates more pain-related disability.
Change in State-Trait Anxiety using the The State-Trait Anxiety Inventory (STAI) | The questionnaire will be done at the baseline (T0), beginning and just after the 20 minutes of application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo) and one week after the last intervention.
  The STAI is a self-report questionnaire used to measure two types of anxiety: state-anxiety (SA) and treatment-anxiety (TA). Each type of anxiety has its own scale of 20 items that are scored. The score for each type of anxiety ranges from 20 to 80. Higher scores indicate greater anxiety.
Change in Patient Global Impression of Change (PGIC) | The questionnaire will be done at the baseline (T0), beginning and just after the 20 minutes of application of each intervention (VR, VR + CN-NINM, VR+CN-NINM placebo) and one week after the last intervention.
  The PGIC is a self-report scale used to measure a person's impression of the effectiveness of a treatment or intervention. It is a 7-point scale on which patients rate their overall change, with scores ranging from "very much improved," to "very much worse".

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Léonard, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement (CdRV), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No